CLINICAL TRIAL: NCT05165407
Title: Sintilimab Combined With IBI310 and Surufatinib for the Treatment of High-grade Advanced-neuroendocrine Neoplasms: a Single Arm, Open-label, Multi Center, Phase II Study
Brief Title: Sintilimab Combined With IBI310 and Surufatinib for the Treatment of G3-NET and NEC (NESSIE)
Acronym: NESSIE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Clinical Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGOG-3006/2021-01
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Neuroendocrine Neoplasm
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — sintilimab; surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab Combined With IBI310 and Surufatinib (Experimental): Surufatinib at a dose of 250mg QD, with Sintilimab injected intravenously 200mg per 3 weeks and IBI310 injected intravenously 1mg/kg per 6 weeks until disease progresses or unacceptable tolerability occurs
  Interventions: Drug: Sintilimab; Drug: IBI310; Drug: Surufatinib

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg will be intravenously administered on Day 1 of each cycle
Drug: IBI310 — IBI310 1mg/kg be intravenously administered on Day 1 of every 2 cycle
Drug: Surufatinib — Surufatinib 250mg will be taken orally once daily continuously
  Other Names: HMPL-012

SUMMARY:
This is a phase II, single arm, open-label, multicenter study to evaluate the efficacy and safety of Sintilimab combined with IBI310 and Surufatinib for the treatment of high-grade advanced-neuroendocrine neoplasm

DETAILED DESCRIPTION:
The study population is about 40 patients with high-grade advanced-neuroendocrine neoplasm, who fails or cannot tolerate standard therapies. Surufatinib 250 mg once a day (QD) will be orally administrated, Sintilimab 200mg will be intravenously administered every 3 weeks and IBI310 1mg/kg will be intravenously administered every 6 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent. For Sintilimab, the upper time limit for treatment is 2 years. The primary objective is objective response rate (ORR) of Sintilimab combined with IBI310 and Surufatinib in patients with advanced high-grade advanced-neuroendocrine neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* Patients who included in this study must fulfil all of the following criteria:

  1. Fully aware of this study and voluntary to sign the informed consent form (the informed consent form must be signed before any trial-specific procedure is performed);
  2. Aged 18-75 (inclusive);
  3. Histologically or cytologically confirmed patients with inoperable or metastatic high-grade neuroendocrine neoplasm (Ki67 index > 20% or with mitotic count of more than 20 mitoses per high power field);
  4. Patients who failed to receive standard treatment (Have progressed on previous treatment, or treatment toxicity and side effects are not tolerated), or cannot receive standard treatment (including patients who are intolerant to standard treatment, who are judged by the investigator to be unsuitable for standard treatment or who refuse to receive standard treatment), or who have no standard treatment plan;
  5. Having clear measurable lesions (according to RECIST 1.1). If the lesion is the only one that has received previous local treatment (radiotherapy, ablation, vascular intervention, etc.), there must be clear imaging evidence of disease progression in that lesion;
  6. Agree to provide tumor specimens (for further diagnosis of pathological grade, detection of PD-L1 expression and lymphocyte infiltration);
  7. ECOG performance status of 0 or 1;
  8. Brain metastases are asymptomatic or stable after local treatment are allowed to be enrolled as long as they meet the following conditions:

  1) Measurable lesions are outside of the central nervous system 2) No central nervous system symptoms or no exacerbation of symptoms for at least 2 weeks 3) No glucocorticoid treatment or discontinuation of glucocorticoid treatment within 7 days before first dose of study treatment.

  9. Patients were allowed to receive palliative radiation therapy, but it ended 14 days before the first dose of study treatment, and the radiation-related toxicity returned to grade 1 or less (CTCAE5.0); 10. Predicted survival ≥ 3 months; 11. Patients with adequate organ functions whose laboratory tests within 7 days before the first dose meet the following requirements:
  1. Absolute neutrophil count (ANC) ≥1.5x109/L within 14 days, without use of granulocyte colony-stimulating factor or other hematopoietic stimulating factor.
  2. Platelet count ≥100×109/L within 14 days, without blood transfusion or use of blood product.
  3. Hemoglobin ≥ 9 g/dL within 14 days, without blood transfusion or erythropoietin.
  4. Total bilirubin ≤1.5 × upper limit of normal (ULN); Such as total bilirubin > 1.5×ULN, but direct bilirubin ≤ ULN was also allowed.
  5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN in patients with liver metastasis).
  6. Serum creatinine ≤1.5×ULN and creatinine clearance rate ≥60 mL /min (calculated according to the Cockcroft-Gault formula).
  7. Good coagulation function, defined as International normalized ratio (INR) or prothrombin time (PT) ≤1.5 ULN;
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can be enrolled; Hypothyroidism that can be controlled only by thyroid hormone replacement therapy can be enrolled;
  9. The myocardial enzyme profile is within the normal range (if the investigator comprehensively determines that the simple laboratory abnormality is not clinically significant, the patients is allowed to be enrolled); 12. Females of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to the first dose (Day 1 of Cycle 1). If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested. All female patients will be considered to be of childbearing potential unless they are naturally postmenopausal, underwent artificial menopause, or are surgically sterile (e.g., hysterectomy, bilateral adnexectomy).

  13. If there is a risk of conception, Male or female patients of childbearing potential volunteer to use effective contraceptive methods (failure rate ≤ 1%) during the study and within 120 days after last administration of the study drug.

Exclusion Criteria:

* Subjects must be excluded from this study when any one of the following criteria is met:

  1. Presence of other malignancies in the past 5 years (except for basal cell carcinoma or squamous cell carcinoma of the skin and carcinoma in situ of the cervix, which were effectively controlled);
  2. Currently participate in an interventional clinical study, or have been treated with another study drug or medical equipment within 4 weeks prior to the first dose;
  3. Previous use of anti (PD-1), anti-PD-L1, anti-PD-L2 or CTLA-4 antibody or any other antibody acting on T cell co-stimulatory or checkpoint pathways (including but not limited to OX-40, CD137, etc.), anti-VEGF/VEGFR-targeted drugs;
  4. Having abnormal thyroid function with symptoms ongoing or requiring treatment at screening (only hypothyroidism that can be controlled by thyroid hormone replacement therapy can be included);
  5. Received systemic therapy with anti-neuroendocrine tumor of proprietary Chinese medicines or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local control of pleural effusion) within 2 weeks prior to the first dose;
  6. Patients with any active autoimmune disorders requiring systematic treatment (e.g., palliative drugs, glucocorticoids, or immunosuppressants) or a history of autoimmune disease in the past 2 years. Alternative therapies (e.g. thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary dysfunction) are not considered systemic;
  7. Use of immunosuppressant within 7 days prior to the first dose, not including local glucocorticoid via nasal spray, inhalation or other routes or systemic glucocorticoid at physiological dose. Note: Physiological doses of glucocorticoids (≤10 mg/ day of prednisone or equivalent dose) are permitted;
  8. Uncontrollable malignant hydrothorax, ascites or pericardial effusion (patients who do not need drainage effusion or who stop drainage for 3 days without significant increase in effusion can be included in the group);
  9. Use of CYP3A potent or moderate inducers during the administration of concomitant medications or within 1 weeks or 5 half-lives (whichever is longer) prior to the first dose (Appendix 3);
  10. Patients who currently have gastric and duodenal active ulcer, ulcerative colitis, or active bleeding in the unresected tumor, or serious gastrointestinal disorders, or other conditions that may cause haemorrhage of digestive tract or perforation;
  11. Patients with evidence or history of obvious bleeding tendency within 2 months prior to the first dose. (bleeding within 2 months > 30 mL, hematemesis, black feces), hemoptysis (within 4 weeks > 5 mL of fresh blood);
  12. Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
  13. A history of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drugs (Sintilimab, IBI310, Surufatinib), or a prior history of severe allergy to any other monoclonal antibody.
  14. Patients with multiple factors affecting oral medication (such as inability to swallow, post-gastrointestinal resection, chronic diarrhea and intestinal obstruction);
  15. Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for hair loss);
  16. Human immunodeficiency virus (HIV) antibody positive;
  17. Untreated active hepatitis B (defined as HBsAg positive with HBV-DNA copy number greater than the upper limit of the normal value in the laboratory department of the research center);

      Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

  1) HBV viral load before initial administration < 1000 copies/mL (200 IU/ml). Subjects should receive anti-HBV therapy to avoid virus reactivation 2) For patients with HBc (+), HBsAg (-), anti-HBS (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but rigorous monitoring of virus reactivation is required;

  18. Patients with known positive hepatitis C virus antibody (HCV Ab) and HCV RNA > 1 × 103 copies/mL;

  19. Vaccination of any live or attenuated live vaccine within 4 weeks prior to the first dose or during the study; Note: Acceptance of injectable inactivated virus vaccine against seasonal influenza is permitted within 30 days prior to first dose; Intranasally administered live attenuated flu vaccines are not allowed;

  20. Pregnant (positive pregnancy test prior to administration) or lactating women;

  21. Presence of any serious or uncontrollable systemic illness;

  22. Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other condition that investigators suspect may prohibit use of the investigational product, affect interpretation of study results, or put the patient at high risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR, RECIST 1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy(up to approximately 2 years)
  The incidence of confirmed complete response or partial response

SECONDARY OUTCOMES:
Objective response rate (ORR, iRECIST 1.1) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy(up to approximately 2 years)
  The incidence of confirmed complete response or partial response
Progression-free Survival (PFS) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anticancer therapy (up to approximately 2 years)
  A duration from the date of initial treatment to disease progression or death of any cause
Duration of response (DoR) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)
  Duration from the first time reported partial response or complete response to the first time of disease progression or death
Overall survival (OS) | From date of first dose of study drug until death caused by any reason (up to approximately 2 years)
  From the time of enrollment to death caused by any reason
Safety of regimen as measured by incidence of adverse events | The safety and tolerability of Surufatinib will be evaluated based on adverse events data. Other safety parameters include physical examination, vital signs, laboratory test results
  From first dose to within 30 days after the last dose
PD-L1 | Up to approximately 2 years
  To evaluate the relationship between the efficacy and tumor biomarkers of PD-L1

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Bejing cancer hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No